CLINICAL TRIAL: NCT04826965
Title: Does Negative Pressure Wound Therapy With Instillation Reduce the Bioburden of Infections of the Upper and Lower Extremity?
Brief Title: VAC Bioburden Wound Care Assessment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Duke University (Other)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00105056
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Results first posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Upper Extremity Wound; Lower Extremity Wound; Soft Tissue Abscesses; Traumatic Wounds

STUDY DESIGN:
Intervention Model Description: Screen 60 subjects in hopes to enroll 40. There will be 20 subjects per arm. All subjects will have a wound vac applied. The randomization will be whether or not irrigation is included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Wound vac application (Active Comparator): Wound vac application for open upper/lower extremity open wound
  Interventions: Device: Wound Vac is applied
- Wound vac application including irrigation (Active Comparator): Wound vac application WITH irrigation for upper/lower extremity open wound
  Interventions: Device: Wound Vac is applied

INTERVENTIONS:
Device: Wound Vac is applied — A wound vac or wound vac with cleanse choice dressing, track pad duo, and saline irrigation is applied.

SUMMARY:
The purpose of this study is to compare the microbiologic burden and need for further operative debridement of patients undergoing primary surgical debridement of infected tissue, soft tissue abscesses, or traumatic wounds of the upper and lower extremity.

DETAILED DESCRIPTION:
Bacterial bio-burden as measured by quantitative microbial PCR prior to debridement, immediately following initial debridement, after 2 days of VAC veraflo (or conventional VAC) therapy, and at the time of repeat operative debridements, if needed. We will use the MicroGen PCR platform (DBA Microgen Diagnostics, LLC, Lubbock, TX.) to report on the bacterial burden (reported on a log scale of bacteria per gram) present at the time of debridement. Our goal is to be able to assess the bioburden quantitatively at each time point to discern a change.

Exploratory outcomes to be measured: number of operative debridements required prior to reconstruction, number of days until final reconstruction, number of days until decision is made by surgeon that further debridements are no longer necessary, length of hospital stay, wound surface area will be monitored from enrollment through when the veraflo is removed. This is likely a 3-month interval.

ELIGIBILITY:
Inclusion Criteria:

* 18+yo with an injury or infection of the upper or lower extremity for which surgical debridement (in the operating room) followed by VAC application is planned.

Exclusion Criteria:

- Patient with wounds distal to the ankle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suhail Mithani, MD, Principal Investigator — Duke Health System
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wound Vac Application | Wound Vac Application Including Irrigation
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wound Vac Application | Wound Vac Application Including Irrigation | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Bio-burden as Measured by Qualitative Microbial PCR (Polymerase Chain Reaction) Prior to First Debridement
Description: Bacterial bio-burden as measured by microbial PCR prior to debridement using the MicroGen PCR platform (DBA Microgen Diagnostics, LLC, Lubbock, TX). Reported as the number of participants with low (< 1x10^5), medium (1x10^5 to 1x10^7), and high (> 1x10^7) counts of bacteria per gram.
Time Frame: Day 1 (day of first operative debridement)
Measure: Count of Participants; unit: Participants
Arm/Group | Wound Vac Application | Wound Vac Application Including Irrigation
Number analyzed (Participants) | 3 | 2
Participants
  Low | 0 | 0
  Medium | 1 | 1
  High | 2 | 1

2. Primary Outcome: Bio-burden as Measured by Qualitative Microbial PCR (Polymerase Chain Reaction) After First Debridement
Description: Bacterial bio-burden as measured by microbial PCR after debridement using the MicroGen PCR platform (DBA Microgen Diagnostics, LLC, Lubbock, TX). Reported as the number of participants with low (< 1x10^5), medium (1x10^5 to 1x10^7), and high (> 1x10^7) counts of bacteria per gram.
Time Frame: Day 1 (day of first operative debridement)
Measure: Count of Participants; unit: Participants
Arm/Group | Wound Vac Application | Wound Vac Application Including Irrigation
Number analyzed (Participants) | 3 | 2
Participants
  Low | 1 | 1
  Medium | 1 | 1
  High | 1 | 0

3. Primary Outcome: Bio-burden as Measured by Qualitative Microbial PCR (Polymerase Chain Reaction) Prior to Second Debridement
Description: as for outcome 1
Time Frame: Day 2 (day of second operative debridement)
Measure: Count of Participants; unit: Participants
Arm/Group | Wound Vac Application | Wound Vac Application Including Irrigation
Number analyzed (Participants) | 3 | 2
Participants
  Low | 1 | 1
  Medium | 1 | 0
  High | 0 | 1
  Not Detected | 1 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Wound Vac Application | Wound Vac Application Including Irrigation
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT04826965/Prot_SAP_000.pdf